CLINICAL TRIAL: NCT00319111
Title: Long-term Open-label Extension Study in Patients With Inoperable Chronic Thromboembolic Pulmonary Hypertension (CTEPH) Who Completed Protocol AC-052-366 (BENEFIT, NCT00313222)
Brief Title: Bosentan in Patients With Inoperable Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Acronym: BENEFIT OL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-370; BENEFIT OL
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; bosentan; BENEFIT; CTEPH; inoperable chronic thromboembolic pulmonary hypertension (CTEPH)
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Bosentan

ARMS (1):
- Bosentan (Experimental): Open label bosentan treatment
  Interventions: Drug: bosentan

INTERVENTIONS:
Drug: bosentan — Oral bosentan
  * Initial dose: 62.5 mg twice a day (b.i.d.) for 4 weeks for all patients
  * Maintenance dose: 125 mg b.i.d. (62.5 mg b.i.d. if weight < 40 kg)

SUMMARY:
The present trial investigates the long-term safety, tolerability and efficacy of bosentan in patients with inoperable CTEPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients having completed the 16-week treatment period of protocol AC-052-366 (NCT00313222)
* Signed informed consent

Exclusion Criteria:

* Any major violation of protocol AC-052-366 (NCT00313222)
* Pregnancy or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 26 centers in 13 countries (Australia, Austria, Belgium, Canada, Czech Republic, France, Germany, Italy, The Netherlands, Poland, Spain, UK, and USA. The first patient started treatment on 26 January 2006 and the last patient received their last dose of study treatment on 23 February 2009.
Pre-assignment Details: In total, 148 of the patients who received randomized treatment in BENEFIT (NCT00313222) rolled over into the BENEFIT OL extension. In addition, 3 patients on bosentan who were prematurely discontinued from BENEFIT (NCT00313222) were also included in the analysis, providing a total of 151 patients
Period: Overall Study
Arm/Group | Bosentan
Started | 151 (148 patients enrolled in BENEFIT OL & 3 prematurely discontinued from BENEFIT (NCT00313222))
Completed | 104
Not Completed | 47
Not completed — Adverse Event | 20
Not completed — Withdrawal of consent | 11
Not completed — Death | 9
Not completed — Lack of clinical improvement | 4
Not completed — Administrative | 2
Not completed — Treatment failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bosentan
Number analyzed (Participants) | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (11.7)
Age, Customized [Number; unit: participants]
  25-81 years | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 51
Region of Enrollment [Number; unit: participants]
  Australia | 17
  Austria | 10
  Belgium | 8
  Canada | 6
  Czech Republic | 20
  France | 18
  Germany | 14
  Italy | 28
  Netherlands | 11
  Poland | 9
  Spain | 3
  United Kingdom | 2
  United States | 5
Six-minute walk test (6MWT) [Mean (Standard Deviation); unit: walk distance (m)] — Exercise capacity was determined for 137 of the 151 participants using the 6MWT. Area used for testing was a minimum of 30m in length and 2-3m in width, with 3m gradations. Areas were well ventilated with air temperature controlled. The test was administered at the same time of day and by the same tester throughout the study. The tester measured the distance walked by non-encouraged patients during the timed 6min period. If the test was stopped before 6 minutes, the main reason for stopping the test was recorded. The tester measured the distance walked by patients during the timed 6min period.
  walk distance (m) | 345.2 (93.4)
Borg dyspnea index [Mean (Standard Deviation); unit: points on a scale] — The Borg dyspnea index was assessed in 136 out of the 151 participants. Maximal dyspnea during the walk test was assessed by the patient using the Borg dyspnea index. Immediately following each walk test, patients rated perceived maximal breathlessness during the walk test on a 12-point scale (0 [nothing at all], 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 [maximum ever experienced]).
  points on a scale | 4.2 (2.2)
World Health Organisation (WHO) functional class [Number; unit: participants] — Disease severity assessed using WHO classification of pulmonary hypertension: Class I: no limitation of physical activity etc.
  Class II: slight limitation of physical activity etc. Class III: marked limitation of physical activity etc. Class IV: inability to carry out physical activity without symptoms. Signs of right heart failure etc.
  WHO functional class was assessed in 139 patients
  participants
    Class I | 3
    Class II | 41
    Class III | 91
    Class IV | 4
    Unassessed | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to All Assessed Time Points in 6-minute Walk Test (6MWT) Distance
Description: Exercise capacity was assessed using the 6MWT. Area used for testing had to be a minimum of 30m in length and 2-3m in width, with 3m gradations. Areas were well ventilated with air temperature controlled. The test was administered at the same time of day and by the same tester throughout the study. The tester measured the distance walked by non-encouraged patients during the timed 6min period. If the test was stopped before 6 minutes, the main reason for stopping the test was recorded. The tester measured the distance walked by patients during the timed 6min period.
Time Frame: Until discontinuation of study drug, up to 3.3 years
Population: Numbers of patients assessed at 6 month, month 12, month 18, month 24 and end of the treatment period were 137, 128, 121, 106, and 137 respectively
Measure: Mean (Standard Deviation); unit: walk distance change from baseline (m)
Arm/Group | Bosentan
Number analyzed (Participants) | 151
walk distance change from baseline (m)
  month 6 | 8.4 (66.4)
  month 12 | 18.2 (64.0)
  month 18 | 17.7 (63.1)
  month 24 | 20.2 (64.8)
  end of the treatment period | 16.9 (69.4)

2. Primary Outcome: Change From Baseline to All Assessed Time Points in Borg Dyspnea Index
Description: Maximal dyspnea during the walk test was assessed by the patient using the Borg dyspnea index. Immediately following each walk test, patients rated perceived maximal breathlessness during the walk test on a 12-point scale (0 [nothing at all], 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 [maximum ever experienced]).
Time Frame: Until discontinuation of study drug, up to 3.3 years
Population: Numbers of patients assessed at 6 month, month 12, month 18, month 24 and end of the treatment period were 136, 127, 120, 105, and 136 respectively
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 151
Scores on a scale
  month 6 | -0.5 (1.7)
  month 12 | -0.4 (1.8)
  month 18 | -0.1 (1.9)
  month 24 | -0.1 (1.9)
  end of the treatment period | -0.2 (2.1)

3. Primary Outcome: Disease Severity - Number of Patients Showing Improvement by One Class or More in World Health Organisation (WHO) Functional Classification of Pulmonary Hypertension (PH)
Description: Disease severity was assessed by WHO classification of PH criteria:
  Class I: no limitation of physical activity (PA). Ordinary PA: no undue dyspnea/fatigue, chest pain, near syncope.
  Class II: slight limitation of PA. Comfortable at rest. Ordinary PA: undue dyspnea/fatigue, chest pain, near syncope.
  Class III: marked limitation of PA. Comfortable at rest. Less than ordinary PA: undue dyspnea/fatigue, chest pain, near syncope.
  Class IV: inability to carry out PA without symptoms. Right heart failure. Dyspnea/fatigue may even have been present at rest. Discomfort increased by any PA.
Time Frame: Until discontinuation of study drug, up to 3.3 years
Population: Numbers of patients assessed at 6 month, month 12, month 18, month 24 and end of the treatment period were 138, 129, 123, 109, and 139 respectively
Measure: Number; unit: participants with improved WHO class
Arm/Group | Bosentan
Number analyzed (Participants) | 151
participants with improved WHO class
  month 6 | 26
  month 12 | 30
  month 18 | 33
  month 24 | 33
  end of treatment period | 30

4. Primary Outcome: Time to Clinical Worsening up to End-of-study
Description: An event of clinical worsening was defined as death during the treatment period, a treatment-emergent adverse event that led to permanent discontinuation of study treatment and with outcome death, hospitalization due to worsening pulmonary hypertension, or lung transplantation. Patients are censored at 1 day after the end of treatment or at day of pulmonary endarterectomy if earlier.
Time Frame: Until discontinuation of study drug, up to 3.3 years
Population: Study population
Measure: Number; unit: participants
Arm/Group | Bosentan
Number analyzed (Participants) | 151
participants
  month 6 (censored) | 11
  month 6 (events) | 8
  month 12 (censored) | 18
  month 12 (events) | 11
  month 18 (censored) | 25
  month 18 (events) | 15
  month 24 (censored) | 34
  month 24 (events)) | 19
  month 30 (censored) | 78
  month 30 (events) | 20
  month 36 (censored) | 122
  month 36 (events) | 21
  end of study (censored) | 130
  end of study (events) | 21

5. Secondary Outcome: Number of Patients With an Adverse Event(s) Leading to Premature Discontinuation of Study Medication
Time Frame: Until discontinuation of study drug, up to 3.3 years
Population: Study population
Measure: Number; unit: participants
Arm/Group | Bosentan
Number analyzed (Participants) | 151
participants | 28

6. Secondary Outcome: Number of Patients Experiencing a Serious Adverse Event(s) up to 28 Days After Study Medication Discontinuation
Time Frame: 28 days after discontinuation of study drug, up to 3.3 years
Population: Study population
Measure: Number; unit: participants
Arm/Group | Bosentan
Number analyzed (Participants) | 151
participants | 51

7. Secondary Outcome: Occurrence of Liver Function Test and Hemoglobin Abnormality
Description: Number of patients with an increase in liver aminotransferases to >3 times upper limit of normal (ULN) or a decrease in hemoglobin concentration to ≤10 g/dL
Time Frame: Until discontinuation of study drug, up to 3.3 years
Population: study population
Measure: Number; unit: participants
Arm/Group | Bosentan
Number analyzed (Participants) | 151
participants
  Increase in liver function test | 27
  Decrease in hemoglobin | 9

ADVERSE EVENTS:
Time Frame: Up to 28 days after the end of study drug
Description: Only treatment emergent adverse events that were serious or lead to premature discontinuation of study treatment were reported during the study. All serious adverse events occurring during and up to 28 days after end-of-study treatment were reported
Arm/Group | Bosentan
Serious Adverse Events (participants affected / at risk) | 51/151
Other Adverse Events (participants affected / at risk) | 11/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan (N=151)
Right ventricular failure (Cardiac disorders) | 11
Cardiac failure (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 3
Chronic right ventricular failure (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 1
Sinoatrial block (Cardiac disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Liver function test abnormal (Investigations) | 5
ECG signs of myocardial ischaemia (Investigations) | 1
Heart rate abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Pneumonia (Infections and infestations) | 2
Catheter related infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 1
Sudden death (General disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Diabetic hyperglycaemic coma (Nervous system disorders) | 1
Alcohol detoxification (Surgical and medical procedures) | 1
Catheterisation cardiac (Surgical and medical procedures) | 1
Lung transplant (Surgical and medical procedures) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Scrotal swelling (Reproductive system and breast disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Temporal arteritis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan (N=151)
HEPATIC ENZYME INCREASED (Investigations) | 3
LIVER FUNCTION TEST ABNORMAL (Investigations) | 3
ANOREXIA (Metabolism and nutrition disorders) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
DYSPEPSIA (Gastrointestinal disorders) | 1
NASAL MUCOSAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from multi-center studies must be published or presented at congresses only in their entirety and not as individual center data, except for ancillary studies. Any study-related article or abstract written independently by investigators should be submitted to Actelion for review at least 60 days prior to submission for publication or presentation.